CLINICAL TRIAL: NCT02577003
Title: A Phase III, Multicenter, Randomized, Placebo-Controlled, Parallel-Group, Double-Blind Trial to Assess the Safety and Efficacy of Addition of Ipragliflozin in Japanese Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Sitagliptin Monotherapy in Addition to Diet and Exercise Therapy
Brief Title: Double-blind Ipragliflozin Add-on Study in Japanese Participants With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Sitagliptin (MK-0431J-843)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431J-843; 153097 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2015-10-14; First posted 2015-10-15 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ipragliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ipragliflozin + Sitagliptin (Experimental): Ipragliflozin once daily for 24 weeks in addition to sitagliptin, diet, and exercise.
  Interventions: Drug: Ipragliflozin; Drug: Sitagliptin
- Placebo + Sitagliptin (Active Comparator): Placebo to ipragliflozin once daily for 24 weeks in addition to sitagliptin, diet, and exercise.
  Interventions: Drug: Placebo; Drug: Sitagliptin

INTERVENTIONS:
Drug: Ipragliflozin — 50 mg tablet administered orally
  Arms: Ipragliflozin + Sitagliptin
Drug: Placebo — Placebo to ipragliflozin tablet administered orally
  Arms: Placebo + Sitagliptin
Drug: Sitagliptin — Background medication; 50 mg tablet administered orally
  Other Names: Januvia®, Tesavel®, Xelevia®, Ristaben®, Glactiv®

SUMMARY:
This is a study to assess the safety and efficacy of the addition of ipragliflozin once daily in Japanese participants with Type 2 diabetes mellitus (T2DM) who have inadequate glycemic control on sitagliptin, diet, and exercise therapy. The primary hypothesis for this study is that the addition of ipragliflozin compared with placebo provides greater reduction in hemoglobin A1C (HbA1c) as assessed by change from baseline at Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Inadequate glycemic control on diet/exercise therapy and sitagliptin monotherapy
* HbA1c ≥7.0% and ≤10.0% before study start

Exclusion Criteria:

* History of Type 1 diabetes mellitus or a history of ketoacidosis
* History of any of the following medications: thiazolidinediones (TZD) and/or insulin within 12 weeks prior to study participation and sodium glucose cotransporter 2 (SGLT2) inhibitors anytime
* Currently has a urinary tract infection or genital infection with subjective symptom

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2015-11-09; Primary Completion 2016-11-25 (Actual); Study Completion 2016-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Kaku K, Kadowaki T, Seino Y, Okamoto T, Shirakawa M, Sato A, O'Neill EA, Engel SS, Kaufman KD. Efficacy and safety of ipragliflozin in Japanese patients with type 2 diabetes and inadequate glycaemic control on sitagliptin. Diabetes Obes Metab. 2021 Sep;23(9):2099-2108. doi: 10.1111/dom.14448. Epub 2021 Jun 15. PMID 34033212

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, all participants received placebo for 2 weeks.
Period: Overall Study
Arm/Group | Ipragliflozin + Sitagliptin | Placebo + Sitagliptin
Started | 73 | 70
Completed | 71 | 65
Not Completed | 2 | 5
Not completed — Adverse Event | 2 | 4
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipragliflozin + Sitagliptin | Placebo + Sitagliptin | Total
Number analyzed (Participants) | 73 | 70 | 143
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.0 (9.1) | 60.0 (10.4) | 60.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 54 | 53 | 107
HbA1c [Mean (Standard Deviation); unit: Percent] | 8.05 (0.83) | 7.99 (0.62) | 8.02 (0.73)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 82.0 (13.5) | 83.4 (16.7) | 82.7 (15.1)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 158.0 (33.2) | 163.0 (26.2) | 160.5 (30.0)
2-hour Post-Meal Glucose (2-hr PMG) [Mean (Standard Deviation); unit: mg/dL] | 225.3 (59.9) | 231.5 (48.9) | 228.3 (54.7)
Glucose Total Area Under the Plasma Concentration Curve from Hour 0 to Hour 2 (AUC0-2hr) after Meal [Mean (Standard Deviation); unit: mg･hr/dL] | 429.4 (86.3) | 443.4 (67.0) | 436.2 (77.5)
Body Weight [Mean (Standard Deviation); unit: kg] | 69.8 (11.7) | 70.1 (11.1) | 69.9 (11.4)
Prior use of other antihyperglycemic agents (AHAs) [Count of Participants; unit: Participants] — Other AHAs refers to the use of AHAs other than sitagliptin within 8 weeks of study start.
  Participants
    Yes | 31 | 30 | 61
    No | 42 | 40 | 82

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 24
Description: HbA1c is measured as percent. Thus, this change from baseline reflects the Week 24 HbA1c percent minus the Week 0 HbA1c percent. Statistical analysis based on a constrained longitudinal data analysis (cLDA) model with terms for treatment, time, prior use of AHAs, the interactions of treatment by time, time by prior use of AHAs, treatment by time by prior use of AHAs, and baseline eGFR value with the constraint that the mean baseline HbA1c is the same for both treatment groups.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of treatment period study medication and have at least one measurement of HbA1c (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Ipragliflozin + Sitagliptin | Placebo + Sitagliptin
Number analyzed (Participants) | 73 | 70
Percent | -0.84 [-0.99 to -0.69] | -0.07 [-0.22 to 0.09]
Statistical Analysis 1: Comparison: Ipragliflozin + Sitagliptin vs Placebo + Sitagliptin; Test type: Superiority; p < 0.001, Constrained longitudinal data analysis; Based on a cLDA model with the terms listed above; Difference in least squares means = -0.77, 95% CI 2-sided [-0.98 to -0.57]

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 26 weeks
Population: All randomized participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Ipragliflozin + Sitagliptin | Placebo + Sitagliptin
Number analyzed (Participants) | 73 | 70
Percentage of participants | 50.7 | 65.7

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 2
Time Frame: Up to 24 weeks
Population: All randomized participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Ipragliflozin + Sitagliptin | Placebo + Sitagliptin
Number analyzed (Participants) | 73 | 70
Percentage of participants | 2.7 | 5.7

4. Secondary Outcome: Change From Baseline in FPG at Week 24
Description: Change from baseline in FPG at Week 24 is defined as Week 24 FPG minus Week 0 FPG. Statistical analysis based on a cLDA model with terms for treatment, time, prior use of AHAs, the interactions of treatment by time, time by prior use of AHAs, treatment by time by prior use of AHAs, and baseline eGFR value with the constraint that the mean baseline FPG is the same for both treatment groups.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of treatment period study medication and have at least one measurement of FPG (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ipragliflozin + Sitagliptin | Placebo + Sitagliptin
Number analyzed (Participants) | 73 | 70
mg/dL | -30.3 [-35.5 to -25.0] | -2.1 [-7.6 to 3.3]
Statistical Analysis 1: Comparison: Ipragliflozin + Sitagliptin vs Placebo + Sitagliptin; Test type: Superiority; p < 0.001, Constrained longitudinal data analysis; Based on a cLDA model with the terms listed above; Difference in least squares means = -28.1, 95% CI 2-sided [-34.8 to -21.5]

5. Secondary Outcome: Change From Baseline in 2-hr PMG at Week 24
Description: Change from baseline in 2-hr PMG at Week 24 is defined as Week 24 2-hr PMG minus Week 0 2-hr PMG. Statistical analysis based on a cLDA model with terms for treatment, time, prior use of AHAs, the interactions of treatment by time, time by prior use of AHAs, treatment by time by prior use of AHAs, and baseline eGFR value with the constraint that the mean baseline 2-hr PMG is the same for both treatment groups.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of treatment period study medication and have at least one measurement of 2-hr PMG (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ipragliflozin + Sitagliptin | Placebo + Sitagliptin
Number analyzed (Participants) | 73 | 70
mg/dL | -52.4 [-61.5 to -43.2] | -3.8 [-13.3 to 5.7]
Statistical Analysis 1: Comparison: Ipragliflozin + Sitagliptin vs Placebo + Sitagliptin; Test type: Superiority; p < 0.001, Constrained longitudinal data analysis; Based on a cLDA model with the terms listed above; Difference in least squares means = -48.5, 95% CI 2-sided [-59.6 to -37.5]

6. Secondary Outcome: Change From Baseline in Glucose Total AUC0-2hr After Meal at Week 24
Description: Change from baseline in glucose total AUC0-2hr after meal at Week 24 is defined as Week 24 glucose total AUC0-2hr after a meal minus Week 0 glucose total AUC0-2hr after a meal. Statistical analysis based on a cLDA model with terms for treatment, time, prior use of AHAs, the interactions of treatment by time, time by prior use of AHAs and treatment by time by prior use of AHAs, and baseline eGFR value with the constraint that the mean baseline glucose total AUC0-2hr after meal is the same for both treatment groups.
Time Frame: Baseline and Week 24 (just before the loading meal [0 min], 30 min, 60 min and 120 min)
Population: All randomized participants who received at least one dose of treatment period study medication and have at least one measurement of glucose total AUC0-2hr after meal (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg･hr/dL
Arm/Group | Ipragliflozin + Sitagliptin | Placebo + Sitagliptin
Number analyzed (Participants) | 73 | 70
mg･hr/dL | -86.9 [-101.0 to -72.9] | -2.3 [-17.0 to 12.3]
Statistical Analysis 1: Comparison: Ipragliflozin + Sitagliptin vs Placebo + Sitagliptin; Test type: Superiority; p < 0.001, Constrained longitudinal data analysis; Based on a cLDA model with the terms listed above; Difference in least squares means = -84.6, 95% CI 2-sided [-102.6 to -66.6]

7. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: Change from baseline in body weight at Week 24 is defined as Week 24 body weight minus Week 0 body weight. Statistical analysis based on a cLDA model with terms for treatment, time, prior use of AHAs, the interactions of treatment by time, time by prior use of AHAs and treatment by time by prior use of AHAs, and baseline eGFR value with the constraint that the mean baseline body weight is the same for both treatment groups.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of treatment period study medication and have at least one measurement of body weight after meal (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Ipragliflozin + Sitagliptin | Placebo + Sitagliptin
Number analyzed (Participants) | 73 | 70
kg | -2.4 [-2.9 to -1.9] | -0.6 [-1.1 to -0.1]
Statistical Analysis 1: Comparison: Ipragliflozin + Sitagliptin vs Placebo + Sitagliptin; Test type: Superiority; p < 0.001, Constrained longitudinal data analysis; Based on a cLDA model with the terms listed above; Difference in least squares means = -1.8, 95% CI 2-sided [-2.5 to -1.1]

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Arm/Group | Ipragliflozin + Sitagliptin | Placebo + Sitagliptin
Serious Adverse Events (participants affected / at risk) | 2/73 | 4/70
Other Adverse Events (participants affected / at risk) | 12/73 | 15/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipragliflozin + Sitagliptin (N=73) | Placebo + Sitagliptin (N=70)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipragliflozin + Sitagliptin (N=73) | Placebo + Sitagliptin (N=70)
Constipation (Gastrointestinal disorders) | 2 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 10 (12) | 10 (12)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.